CLINICAL TRIAL: NCT04283474
Title: A Phase 1, Single-Blind, Placebo-Controlled, Single and Multiple Ascending Dose Study to Assess the Safety, Tolerability, and Pharmacokinetics of XG005-03 (Topical) in Healthy Subjects
Brief Title: Phase 1 XG005-03 Topical Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Xgene Pharmaceutical Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Basic Science
Other Study IDs: PR-XG005-03-PK-01
Record Dates: First submitted 2020-02-12; First posted 2020-02-25 (Actual); Last update posted 2021-03-25 (Actual); Status verified 2021-03

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- XG005-03 (Experimental): XG005-03 in 3 dose levels
  Interventions: Drug: XG005-03
- Placebo (Placebo Comparator): Placebo in all cohort
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: XG005-03 — 3 different concentrations (1%, 5%, 10%) of XG005-03 topical formulation
  Arms: XG005-03
Drug: Placebo — Placebo topical formulation
  Arms: Placebo

SUMMARY:
Phase 1, randomized, single-blinded, placebo-control, ascending single and multiple dose of the PK, safety, and tolerability of XG005-03 topical formulation in Healthy Volunteers.

DETAILED DESCRIPTION:
This is a single-blind, placebo-controlled study which will investigate the PK, safety and tolerability of XG005-03 topical formulation, in three ascending concentrations after single and multiple topical applications in healthy subjects. The trial consists of two parts: a single ascending dose (SAD; Part 1) and a multiple ascending dose (MAD; Part 2). The MAD study will begin after the SAD portion of the study is complete.

The study will consist of 4 weeks of screening period, treatment period (1 day of dosing for SAD and 6.5 days for MAD), and 14 days of safety follow-up period. Each subject will serve as his/her own control, as the XG005-03 and placebo will be applied on contralateral legs. Application of XG005-03 or placebo to a particular leg will be randomly assigned.

Approximately 36 healthy subjects will be enrolled. Eighteen healthy subjects (3 alternates per dose group) in Part 1 (SAD) and Part 2 (MAD), who fulfill eligibility criteria will receive the study drug: XG005-03 (1%, 5%, and 10%) and placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males or females between 18 and 55 years of age
2. BMI 18.0 to 30.0 kg/m2
3. Non-pregnant, non-breastfeeding female subjects

Exclusion Criteria:

1. Unstable or severe illness
2. Skin infection or lesion
3. Subjects with scars, moles, tattoos at application site
4. Expose to excessive UV
5. Hypersensitivity or allergy to NSAID

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2020-02-28 (Actual); Primary Completion 2021-01-28 (Actual); Study Completion 2021-01-28 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic Analyses | Day 1 to 4 days after last dose
  peak concentration (Cmax)
Pharmacokinetic Analyses | Day 1 to 4 days after last dose
  time to peak concentration (Tmax)
Pharmacokinetic Analyses | Day 1 to 4 days after last dose
  terminal elimination rate constant (Kel)
Pharmacokinetic of XG005-03 in 1%, 5%, and 10% concentrations | Day 1 to 4 days after last dose
  half-life (t½)
Pharmacokinetic Analyses | Day 1 to 4 days after last dose
  area under the concentration-time curve from time 0 to the last measurable concentration timepoint (AUC0-t)
Pharmacokinetic Analyses | Day 1 to 4 days after last dose
  area under the concentration-time curve, extrapolated to infinity (AUC0-∞)

SECONDARY OUTCOMES:
Safety Analyses | treatment to follow up period, a average 20 days
  Adverse Event
Safety Analyses | treatment to follow up period, a average 20 days
  ECG-heart rate
Safety Analyses | treatment to follow up period, a average 20 days
  ECG-PR
Safety Analyses | treatment to follow up period, a average 20 days
  ECG-QRS
Safety Analyses | treatment to follow up period, a average 20 days
  ECG-QT
Safety Analyses | treatment to follow up period, a average 20 days
  ECG-QTc
Safety Analyses | treatment to follow up period, a average 20 days
  Skin Assessment Grading-Burger and Bowman scale
Safety Analyses | treatment to follow up period, a average 20 days
  Vital Sign-Systolic Blood Pressure
Safety Analyses | treatment to follow up period, a average 20 days
  Vital Sign-Diastolic Blood Pressure
Safety Analyses | treatment to follow up period, a average 20 days
  Vital Sign-Pulse Rate
Safety Analyses | treatment to follow up period, a average 20 days
  Vital Sign-Tympanic Temperature
Safety Analyses | treatment to follow up period, a average 20 days
  Vital Sign-Respiratory Rate

CONTACTS AND LOCATIONS:
Overall Officials: Feng Xu, PHD, Study Chair — Xgene Pharmaceutical Group
Locations (1):
- CMAX Clinical Research Pty Ltd, Adelaide, South Australia, Australia

IPD SHARING:
Plan to Share IPD: No